CLINICAL TRIAL: NCT03870009
Title: Validation of a Semi-automatized Method to Detect Cyclic Hyperinflation on CT-scan in ARDS
Acronym: CT4-ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL18_1001; 2019-A00024-53 (Other: ANSM)
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2022-08

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: ARDS; computed tomography; cyclic hyperinflation; mechanical ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARDS patients (Experimental): All the patients will be evaluated with the same procedure, as the study relates to evaluation of the diagnostic performance of a semi-automated method to detect cyclic hyperinflation on CT scan
  Interventions: Other: ARDS patients

INTERVENTIONS:
Other: ARDS patients — The patient will be installed on the scanner bed. Two series of tomographic sections will be acquired: one during an expiratory break, the other during an inspiratory pause.
  cyclic hyperinflation measured by semi-automatic segmentation and by manual segmentation
  Other Names: CT measurements

SUMMARY:
This study aims to validate a semi-automatized method to quantify cyclic hyperinflation on CT-scan of ARDS patients.

The gold standard will be cyclic hyperinflation assessed on the same CT scan, using manual segmentation of the lung.

ELIGIBILITY:
Inclusion Criteria:

* ARDS patients defined by the Berlin definition
* invasive mechanical ventilation with an arterial oxygen pressure (PaO2)/inspired fraction of oxygen (FiO2) ratio ≤ 200 mm Hg
* Indication of CT scan identified by the clinician in charge
* oesophageal catheter already inserted

Exclusion Criteria:

* requirement of contrast agent for a chest CT-scan
* ARDS criteria present for more than 72 hours
* Chronic Obstructive Pulmonary Disease (COPD) on a previous lung function test
* pneumothorax or bronchopleural fistula
* patient without both sedation and neuromuscular blocking agents
* contra-indication to transport to the imaging facility
* treatment with extracorporeal membrane oxygenation or extracorporeal carbon dioxide (CO2) removal
* Latex or curare allergy
* patient previously included in the study
* pregnancy
* patient under limitation of care
* patient under an exclusion period following inclusion in another clinical trial
* patient under a legal protective measure
* patient unaffiliated with social security
* inform consent not obtained by next of kin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
cyclic hyperinflation measured by manual segmentation | 2 hours after inclusion
  Bias and precision of semi-automated measure will be assessed with the Bland and Altman Technique, using cyclic hyperinflation by manual segmentation as a reference
cyclic hyperinflation measured by semi-automated segmentation | 2 hours after inclusion
  Bias and precision of semi-automated measure will be assessed with the Bland and Altman Technique, using cyclic hyperinflation by manual segmentation as a reference

SECONDARY OUTCOMES:
prevalence of cyclic hyperinflation on CT scan | 2 hours after inclusion
  cyclic hyperinflation assessed by manual segmentation on CT scan
area under receiver operating characteristic (ROC) curve of respiratory system driving pressure to detect cyclic hyperinflation assessed by manual segmentation | 2 hours after inclusion
area under ROC curve of transpulmonary driving pressure to detect cyclic hyperinflation assessed by manual segmentation | 2 hours after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jean Christophe Richard, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Croix Rousse Hospital, Lyon, France

REFERENCES:
- [Result] E. Dávila Serrano, François Dhelft, Laurent Bitker, Jean-Christophe Richard, Maciej Orkisz. Software for CT-image Analysis to Assist the Choice of Mechanical-ventilation Settings in Acute Respiratory Distress Syndrome. 2020 International Conference on Computer Vision and Graphics (ICCVG 2020), Sep 2020, Varsovie, Poland. ff10.1007/978-3-030-59006-2_5ff. ffhal-02887264